CLINICAL TRIAL: NCT04616248
Title: A Phase I Study of In Situ Immunomodulation With CDX-301, Radiotherapy, CDX-1140, and Poly-ICLC in Patients With Unresectable and Metastatic Solid Tumors With Injectable Palpable Disease
Brief Title: In Situ Immunomodulation With CDX-301, Radiation Therapy, CDX-1140 and Poly-ICLC in Patients w/ Unresectable and Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1B-22-2; NCI-2022-07303 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1B-22-2 (Other: University of Southern California)
Record Dates: First submitted 2020-10-26; First posted 2020-11-04 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Prognostic Stage IV Breast Cancer AJCC v8; Unresectable Breast Carcinoma; Metastatic Melanoma; Unresectable Melanoma; Cutaneous Squamous Cell Carcinoma; Merkel Cell Carcinoma; Soft Tissue Sarcoma; Bone Sarcoma; Sarcoma,Soft Tissue; Sarcoma of Bone; Basal Cell Carcinoma
Keywords: High-grade bone sarcoma; High-grade soft tissue sarcoma; Basal Cell Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Melanoma; Carcinoma, Merkel Cell; Sarcoma; Bone Neoplasms; Osteosarcoma; Carcinoma, Basal Cell | interventions — poly ICLC; Radiotherapy; Radiation; flt3 ligand protein; pembrolizumab; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort A (immunomodulators, radiation therapy) (Experimental): Patients receive recombinant Flt3 ligand IT on days 1-5 and undergo radiation therapy on day 8 or 9. Patients also receive agonistic anti-CD40 monoclonal antibody CDX-1140 IT and Poly-ICLC IT on day 9 or 10. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anti-CD40 Agonist Monoclonal Antibody CDX-1140; Drug: Poly ICLC; Radiation: Radiation Therapy; Biological: Recombinant Flt3 Ligand
- Cohort B (immunomodulators, radiation therapy) (Experimental): Patients receive recombinant Flt3 ligand IT on days 1-5 and also receive pembrolizumab (IV), tocilizumab (SC) as well as undergo radiation therapy on day 8 or 9. Patients also receive agonistic anti-CD40 monoclonal antibody IT and IV over 90 minutes and Poly-ICLC IT on day 9 or 10. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anti-CD40 Agonist Monoclonal Antibody CDX-1140; Drug: Poly ICLC; Radiation: Radiation Therapy; Biological: Recombinant Flt3 Ligand; Drug: Pembrolizumab; Drug: Tocilizumab

INTERVENTIONS:
Biological: Anti-CD40 Agonist Monoclonal Antibody CDX-1140 — Given IT
  Other Names: Agonist CD40 Antibody CDX-1140; Anti-CD40 Agonistic Monoclonal Antibody CDX-1140; CDX 1140; CDX-1140
Drug: Poly ICLC — Given IT
  Other Names: Hiltonol; Poly I:Poly C with Poly-L-Lysine Stabilizer; poly-ICLC; PolyI:PolyC with Poly-L-Lysine Stabilizer; Polyinosinic-Polycytidylic Acid Stabilized with Polylysine and Carboxymethylcellulose; Polyriboinosinic-Polyribocytidylic Acid-Polylysine Carboxymethylcellulose; Stabilized Polyriboinosinic/Polyribocytidylic Acid
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Biological: Recombinant Flt3 Ligand — Given IT
  Other Names: CDX-301; FLT 3 Ligand; FLT3 Ligand; Flt3-Ligand; Flt3L; Mobist; Mobista; rhuFlt3L
Drug: Pembrolizumab — Given IV
  Other Names: Keytruda
  Arms: Cohort B (immunomodulators, radiation therapy)
Drug: Tocilizumab — Given SC
  Other Names: Actemra
  Arms: Cohort B (immunomodulators, radiation therapy)

SUMMARY:
This phase I trial evaluates the safety and effectiveness of in situ immunomodulation with CDX-301, radiotherapy, CDX-1140 and Poly-ICLC (Cohort A) and these with intravenous (IV) pembrolizumab and subcutaneous (SC) tocilizumab (Cohort B) in treating patients with unresectable and measurable metastatic melanoma, cutaneous squamous cell carcinoma (SCC), basal cell carcinoma (BCC), Merkel cell carcinoma, high-grade bone and soft tissue sarcoma or HER2/neu(-) breast cancer. CDX-301 may induce cross-presenting dendritic cells, master regulators in the immune system. Radiation therapy uses high energy to kill tumor cells and release antigens that may be picked up, processed and presented by cross-presenting dendritic cells. CDX-1140 and Poly-ICLC may activate tumor antigen-loaded,cross-presenting dendritic cells, and generate tumor-specific T lymphocytes, a type of immune cells, that can search out and attack cancers. Giving immune modulators and radiation therapy may stimulate tumor cell death and activate the immune system.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety profile of in situ immunomodulation with CDX-301, radiotherapy, CDX-1140, and Poly-ICLC (Cohort A) and these with pembrolizumab (IV) and tocilizumab (SC) (Cohort B) in unresectable and metastatic melanoma, cutaneous squamous cell carcinoma, basal cell carcinoma, Merkel cell carcinoma, high-grade bone and soft tissue sarcoma or breast cancer patients with injectable palpable disease by determining the maximum tolerated dose (MTD) of CDX-1140 that has an acceptable adverse event profile.

SECONDARY OBJECTIVE:

I. To evaluate the immune signatures in the tumor microenvironment before and after in situ immunomodulation with CDX-301, radiotherapy, CDX-1140, and Poly-ICLC (Cohort A) and these with pembrolizumab (IV) and tocilizumab (SC) (Cohort B).

EXPLORATORY OBJECTIVES:

I. To record the overall response rate (ORR) (complete response [CR] and partial response [PR]) of injected as well as distant uninjected metastatic lesions in metastatic melanoma, cutaneous SCC, basal cell carcinoma, Merkel cell carcinoma, high-grade bone and soft tissue sarcoma or breast cancer patients with injectable palpable disease treated with in situ immunomodulation with CDX-301, radiotherapy, CDX-1140, and Poly-ICLC (Cohort A) and these with pembrolizumab (IV) and tocilizumab (SC) (Cohort B) by immune-related Response Evaluation Criteria In Solid Tumors (irRECIST) response assessment.

II. To record the overall survival (OS) and progression free survival (PFS) in unresectable and metastatic melanoma, cutaneous SCC, basal cell carcinoma, Merkel cell carcinoma, high-grade bone and soft tissue sarcoma or breast cancer patients with injectable palpable disease treated with in situ immunomodulation with CDX-301, radiotherapy, CDX-1140, and Poly-ICLC (Cohort A) and these with pembrolizumab (IV) and tocilizumab (SC) (Cohort B).

III. Examine changes in the levels of T-cell subsets/myeloid derived suppressor cells (MDSC)/cytokines in peripheral blood (PB) of unresectable and metastatic melanoma, cutaneous SCC, basal cell carcinoma, Merkel cell carcinoma, high-grade bone and soft tissue sarcoma or breast cancer patients with injectable palpable disease treated with in situ immunomodulation with CDX-301, radiotherapy, CDX-1140, and Poly-ICLC (Cohort A) and these with pembrolizumab (IV) and tocilizumab (SC) (Cohort B).

OUTLINE:Cohort A will evaluate safety of intratumoral administration of CDX-1140 in combination with CDX-301, radiotherapy and Poly-ICLC. Once cohort A is finished, patients will be enrolled to cohort B to evaluate safety of intratumoral + intravenous administration of CDX-1140 in combination with CDX-301, radiotherapy, pembrolizumab, tocilizumab, and Poly-ICLC.

COHORT A: Patients receive recombinant Flt3 ligand intratumorally (IT) on days 1-5 and agonistic anti-CD40 monoclonal antibody CDX-1140 IT with Poly-ICLC IT on day 9 or 10. Patients also undergo radiation therapy on day 8 or 9. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

COHORT B: Patients receive recombinant Flt3 ligand IT on days 1-5 and agonistic anti-CD40 monoclonal antibody CDX-1140 IT and intravenously (IV) over 90 minutes with Poly-ICLC IT on day 9 or 10. Patients also receive pembrolizumab (IV), tocilizumab (SC), as well as undergo radiation therapy on day 8 or 9. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3-6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Have clinically or pathologically confirmed diagnosis of unresectable and metastatic melanoma, cutaneous SCC, basal cell carcinoma, Merkel cell carcinoma, high-grade bone and soft tissue sarcoma or HER2/neu (-) breast cancer with no curative treatment options.
* The unresectable disease to be irradiated and injected with medications must be located in breast, dermal, subcutaneous, or soft tissue, or lymph nodes with the longest axis of the tumor 2-7 centimeters, and should be considered safe for injection by the investigator.
* The metastatic disease must be measured per irRECIST criteria.
* Patient must have lesion that can be biopsied and is willing to undergo the procedure as part of the protocol.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 1.
* Participants of child-bearing potential and men must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* For patients with history of radiotherapy to the same location that will be treated on study, he/she will be eligible only if the prior radiation dose was under or equal to 68 Gy total and delivered more than 6 months prior to planned re-treatment. (The cumulative dose received to the irradiated area will be no more than 87 Gy total, including a maximum of 68 Gy allowed from prior treatment course.)
* Patient requires the use of radiation therapy to the target lesion of palliation of symptoms and/or achieving local control as part of standard of care as deemed appropriate by treating radiation oncologist.
* Patients must agree to radiation to the tumor.
* Any line of therapy allowed, radiologically or clinically confirmed progression on prior therapy
* Must have adequate organ and marrow function present as defined below:

  * Platelets >= 100,000/uL
  * Hemoglobin >= 8.0 g/dL
  * Absolute neutrophil count (ANC) >= 1500/uL
  * Total bilirubin =< 1.5 X institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional ULN.
  * Creatinine =< 1.5 X ULN OR creatinine clearance >= 50 mL/min per Cockcroft-Gault equation for patients with creatinine levels greater than ULN.
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.
* Patients must agree to injections of CDX-301, CDX-1140, and poly-ICLC.
* Patients must agree to appropriate clinical monitoring to receive the study regimens.
* Patients must agree to photos of tumors and use of the photos for publication.
* Patients should have an administration site for all injections that is free of potentially complicating dermatologic conditions such as rashes.

Exclusion Criteria:

* Patients currently treated with systemic immunosuppressive agents, including steroids, are ineligible until 3 weeks after removal from immunosuppressive treatment. (inhaled steroids are allowed)
* Patients with HER2+ breast cancer
* Concurrent use of targeted therapy including CDK4/6, mTOR, PIK3CA, PARP, BRAF, MEK, hedgehog inhibitors or chemotherapy (endocrine therapy is allowed).
* Targeted therapy including CDK4/6, mTOR, PIK3CA, PARP, BRAF, MEK, hedgehog inhibitors, chemotherapy, or immunotherapy within 2 weeks prior to first dosing of study agent. (endocrine therapy is allowed).
* Patients with active or history of autoimmune disease or history of transplantation except for the patients with Graves' disease with ablative therapy of total thyroidectomy.
* Patients with history of (non-infectious) pneumonitis/interstitial lung disease, including grade 1 pneumonitis (asymptomatic; clinical or diagnostic observations only; intervention not indicated).
* Patients with prior history of acute myeloid leukemia (AML) or known FLT3 aberrations
* Pregnant or nursing female participants.
* Unwilling or unable to follow protocol requirements.
* Patients with known serious mood disorders. (Major depression diagnosis is an exclusion: Other stable mood disorders on stable therapy for > 6 months or not requiring therapy may be allowed after consultation with principal investigator [PI]).
* Cardiac risk factors including:

  * Patients experiencing cardiac event(s) (acute coronary syndrome, myocardial infarction, or ischemia) within 3 months of signing consent.
  * Patients with a New York Heart Association classification of III or IV.
* Patients with uveal melanoma.
* Patients with uncontrolled diseases other than cancer may be excluded if after consultation with PI and research team it is decided it might affect the treatment efficacy or toxicity.
* Evidence of current drug or alcohol abuse or psychiatric impairment, which in the investigator's opinion will prevent completion of the protocol therapy or follow-up. Specific testing is not required, however may be done as clinically indicated.
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug.
* Participants with symptomatic known brain metastases < 4 weeks from radiation treatment should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Other invasive cancers diagnosed < 3 years back that required systemic treatment. If diagnosed with other invasive cancer >= 3 years, should have complete recovery from all systemic toxicity except neuropathy, vitiligo, alopecia, and endocrinopathies on stable hormone replacement therapy.
* Live vaccines within 30 days prior to the first dose of trial treatment and while participating in the trial. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine.
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected).
* Current use of anticoagulants (warfarin, heparin) at therapeutic levels.
* Patients who have had stroke/TIA and DVT/PE within the last 12 months.
* Patients at risk for impending visceral crisis of the liver and lungs as follows, or any condition which in the patient's primary treating oncologist's opinion deems the participant an unsuitable candidate to receive study drug:

  * A visceral crisis of the liver exists when bilirubin levels increase very rapidly (>1.5 times the upper limit of normal) without the presence of Gilbert syndrome (i.e., Meulengracht syndrome) or a biliary tract obstruction.
  * A visceral crisis of the lungs can be assumed when dyspnea at rest increases more rapidly and cannot be relieved by pleural drainage.
* Radiation induced angiosarcoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2027-01-09 (Estimated); Study Completion 2028-01-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days
Maximum tolerated dose or maximum administered dose | Up to 30 days
  The dose limiting toxicity rate will be estimated by cohort and dose-level (if appropriate) using 90% confidence intervals obtained by Jeffrey's prior method.

SECONDARY OUTCOMES:
Changes in Immune signatures in the tumor microenvironment | Baseline up to 2 years
  Will examine changes in the immune biomarkers levels from baseline to end of treatment
Changes in the levels of infiltrating CD4+ and CD8+ T cells | Baseline up to 2 years
  Will examine changes in the levels of infiltrating CD4+ and CD8+ T cells and their proteomic, genomic and transcriptomic signatures in the tumor microenvironment. The immune biomarker levels are treated as continuous variables and will be summarized in the overall sample and within treatment-arm by time-point using the mean and standard error, and graphically using dot-plots.
Changes in the levels of infiltrating myeloid cell subsets | Baseline up to 2 years
  Will examine changes in the levels of infiltrating myeloid cell subsets including dendritic cells (DCs), macrophages, and monocytes, and their proteomic, genomic and transcriptomic signatures in the tumor microenvironment. The immune biomarker levels are treated as continuous variables and will be summarized in the overall sample and within treatment-arm by time-point using the mean and standard error, and graphically using dot-plots.
Changes in the levels of PD-L1 expression | Baseline up to 2 years
  Will examine changes in the levels of PD-L1 expression within both neoplastic and nonneoplastic stromal elements of the tumor microenvironment. The immune biomarker levels are treated as continuous variables and will be summarized in the overall sample and within treatment-arm by time-point using the mean and standard error, and graphically using dot-plots.

OTHER OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  ORR of distant uninjected metastatic lesions is defined as partial or complete response within 6 months of initiating combination therapy. Overall response will be summarized overall and by cohort using frequencies and relative frequencies, where the overall response rate will be estimated using a 90% confidence interval obtained by Jeffrey's prior method.
Overall survival | From treatment initiation until death due to any cause (event) or last follow-up, assessed up to 2 years
  Will be summarized in the overall sample and by cohort using standard Kaplan-Meier methods; where estimates of the median will be obtained with 90% confidence intervals.
Progression free survival | From treatment initiation until disease progression, death due to disease (events), or last follow-up, assessed at 1 year
  Will be summarized in the overall sample and by cohort using standard Kaplan-Meier methods; where estimates of the median will be obtained with 90% confidence intervals.
Changes in the levels of peripheral blood (PB) biomarkers | Baseline up to 2 years
  Will examine changes in the levels of PB biomarkers such as T-cell subsets/myeloid derived suppressor cells (MDSC)/cytokines in metastatic breast cancer patients treated with in situ immunomodulation with CDX-301, radiotherapy, CDX-1140, and poly-ICLC.

CONTACTS AND LOCATIONS:
Overall Officials: Fumito Ito, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California